CLINICAL TRIAL: NCT01273363
Title: Non-interventional Retrospective Multicenter Study of Patients With Bronchial Asthma During a Routine Visit to Out of Patients' Clinics
Acronym: NIKA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RRU-DUM-2010/1
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: Asthma; Asthma in Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Male and female over 18. Patients with asthma diagnosed in accordance with the Global Initiative for Asthma within 6 months before inclusion into the study and without changes in treatment for 2 months before inclusion

SUMMARY:
To assess asthma control in Russian patients according to the new criteria provided in the international guidelines and identify pharmacological approaches that provide a higher level of overall asthma control

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over 18 years of age
* Patients with asthma diagnosed in accordance with the Global Initiative for Asthma (GINA [xv]) within 6 months before inclusion into the study. Patients with no changes in their treatment within 2 months before inclusion into the study
* Patients who signed their informed consents to collection and further processing of data on their disease course

Exclusion Criteria:

* Asthma patients with an exacerbation at the moment of inclusion.
* Patients on β-blockers.
* Patients with COPD, mucoviscidosis or bronchiectasis, Severe heart failure (NYHA functional class III-IV), Renal insufficiency, Cancer, Previous stroke.
* Pregnant women.
* Patients following a major surgery, Hepatic insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To assess asthma control in Russian patients acc. to the new criteria in the international guidelines (Standardizing Endpoints for Clinical Asthma Trials and Clinical Practice) and identify pharmacological approaches provided a higher level of control | 1 visit for 3 month

SECONDARY OUTCOMES:
To determine the main demographic, clinical and pharmacoepidemiological characteristics of low-control patients. | 1 visit for 3 month
To assess comparative value of the Asthma Control Questionnaire (ACT) and Asthma Control Questionnaire (ACQ) with regard to their use in clinical practice in Russia | 1 visit for 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Stepanov, Prof., Study Director — AstraZeneca
Locations (12):
- Russia (12):
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, N.Novgorod
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Yekaterinburg